CLINICAL TRIAL: NCT06005207
Title: A Single-center Randomized Controlled Trial of Vaginal Progesterone to Improve Clinical Pregnancy Outcomes in Patients With Repeated Implantation Failure
Brief Title: Vaginal Progesterone Improves Clinical Outcomes of RIF Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, principal investigator, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ-RIF-P-2023
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal progesterone supplementation (Experimental): 90 mg progesterone vaginal sustained-release gel is added daily to induce endometrial transformation and luteal support
  Interventions: Drug: progesterone vaginal sustained-release gel
- Regular progesterone (No Intervention): No additional vaginal progesterone gel, routine endometrial transformation and luteal support drugs

INTERVENTIONS:
Drug: progesterone vaginal sustained-release gel — 90 mg progesterone vaginal sustained-release gel is added daily during endometrial transformation and luteal support
  Arms: Vaginal progesterone supplementation

SUMMARY:
This study is a single-center, randomized, controlled prospective study. Those patients with repeated implantation failure (RIF) who will recieve frozen thawed embryo transfer (FET) are enrolled in the study. To determine the effect of vaginal progesterone on the clinical pregnancy outcomes of RIF patients.

DETAILED DESCRIPTION:
According to the enrollment and exclusion criteria, the patients were enrolled, and the subjects were randomly divided into two groups by computer randomization. Group A was the vaginal progesterone added group (test group). Group B was the regular FET group (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 20 and 40 years old;
2. BMI: 18-28 kg/m2；
3. Consistent with the diagnosis of repeated implantation failure of unknown reasons, the previous embryo transfer situation meets one of the following:

   Total embryos transferred ≥ 4 high-quality cleavage-stage embryos; ≥ 2 blastocysts; ≥ 2 high quality cleavage-stage embryos +≥ 1 blastocysts;
4. At least 1 high-quality embryo remained for embryo transfer;
5. Volunteer to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Patients with recurrent pregnancy loss (≥ 2 biochemical pregnancies or ≥ 2 spontaneous abortions);
2. Adverse pregnancy history (stillbirth, fetal malformation, etc.);
3. Severe paternal factors: need for TESA or PESA;
4. PGT;
5. Failure of embryo implantation due to any definite reason, including but not limited to: endometrial adhesion (moderate to severe), thin endometrium (<7 mm before transformation), endometritis, endometriosis (medium or severe), adenomyosis, untreated hydrosalpinx, hysteromyoma (submucosal fibroids, non submucosal fibroids > 4.0 cm and/or endometrial compression), reproductive malformation, serious immune disease, serious coagulation function abnormality;
6. Chromosome abnormality of either spouse;
7. Those with contraindications to pregnancy or assisted reproductive technology.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Embryo implantation rate | 45 days after embryo transfer
  The proportion of the number of implanted embryos to the total number of transferred embryos is the embryo implantation rate.

SECONDARY OUTCOMES:
Clinical pregnancy rate | 45 days after embryo transfer
  Clinical pregnancy is defined as the presence of gestational sac observed by ultrasound. The proportion of clinical pregnancy cycles to total FET cycles is the clinical pregnancy rate.
Early pregnancy loss rate | 12 weeks after embryo transfer
  The early pregnancy loss rate refers to the proportion of patients with pregnancy loss before 12 weeks of gestation in the total clinical pregnancy patients.
Persistent pregnancy rate | 20 weeks after embryo transfer
  The ratio of the number of pregnancies lasting to 20 weeks to the number of transplant cycles.
Live birth rate | 40 weeks after embryo transfer
  The ratio of the number of live fetal delivery cycles to the number of transplantation cycles after 28 weeks of pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China